CLINICAL TRIAL: NCT01196637
Title: Thoracic Outlet Syndrome: Case Reports and Analysis - Ultrasound Imaging and Pathomechanics of Brachial Plexus Compression
Brief Title: Thoracic Outlet Syndrome: Case Reports and Analysis With Ultrasound Imaging
Status: Completed | Type: Observational
Sponsor: EMG Labs of Arizona Arthritis & Rheumatology Associates (Other)
Responsible Party: Benjamin M. Sucher, D.O. / Medical Director, EMG Labs of AARA
Other Study IDs: TOS-US BP JAOA
Record Dates: First submitted 2010-09-05; First posted 2010-09-08 (Estimated); Last update posted 2010-09-09 (Estimated); Status verified 2010-09

CONDITIONS: Thoracic Outlet Syndrome
Keywords: thoracic outlet syndrome; brachial plexopathy; ultrasonography
MeSH Terms: conditions — Thoracic Outlet Syndrome; Brachial Plexus Neuropathies

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Thoracic outlet syndrome: These patients have documented thoracic outlet syndrome
- Normal Subjects: These patients have no thoracic outlet syndrome

SUMMARY:
Thoracic outlet syndrome is caused by compression of the brachial plexus, in most cases under the pectoralis minor muscle in the infraclavicular region of the shoulder. The hypothesis is that ultrasound imaging can be used to visualize brachial plexus compression and distortion of the pectoralis muscle during arm activity, such as abduction, and that normal subjects will not demonstrate any plexus compression or muscle distortion.

DETAILED DESCRIPTION:
Four patients with thoracic outlet syndrome (TOS) underwent clinical exam and nerve testing to prove that they had TOS and no other nerve abnormality. They subsequently had ultrasound imaging of the shoulder (infraclavicular region) at rest and during arm abduction stress testing. Two control subjects had similar clinical exams and nerve testing to prove they did not have TOS, and then underwent similar ultrasound stress testing. The TOS patients demonstrated brachial plexus compression and pectoralis minor muscle distortion during the stress tests, and the normal subjects showed no plexus compression or muscle distortion.

ELIGIBILITY:
INCLUSION CRITERIA:

Thoracic outlet patients must have:

* symptoms consistent with thoracic outlet syndrome, and
* no electrical testing abnormality, and
* positive arm abduction stress tests.

Normal subjects must have:

* no upper limb symptoms, or
* normal nerve testing, and
* negative arm abduction stress test

EXCLUSION CRITERIA:

Thoracic outlet patients excluded if they have:

* nerve test abnormalities, or
* negative arm abduction stress test

Normals excluded if they have:

* abnormalities on nerve testing, or
* positive arm abduction stress tests

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients with upper limb symptoms of pain, numbness, tingling, or weakness, aggravated by arm abduction; Adult patients with no upper limb symptoms
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2010-06; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Brachial plexus compression on ultrasound imaging in thoracic outlet syndrome patients | 4 months

SECONDARY OUTCOMES:
No brachial plexus compression in normal subjects | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin M Sucher, D.O., Principal Investigator — EMG Labs of AARA
Locations (1):
- EMG Labs of AARA, Paradise Valley, Arizona, United States